CLINICAL TRIAL: NCT04383314
Title: A Longitudinal, Single-center Study Investigating the Effects of Exercise on Hyaluronan Accumulation in Skeletal Muscle in Individuals With Type 2 Diabetes Mellitus
Brief Title: Targeting Hyaluronan Accumulation Through Exercise in T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-01913
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Program Group (Experimental): Participants will be prescribed an individualized 10-week exercise program with both aerobic and resistance components, based on the American College of Sports Medicine (ACSM) Guidelines.
  Interventions: Behavioral: 10-week exercise program on HA accumulation

INTERVENTIONS:
Behavioral: 10-week exercise program on HA accumulation — A 10-week exercise program with both aerobic and resistance components, based on the American College of Sports Medicine (2010), will be individually prescribed to 25 T2DM patients.Exercise training will be performed on Days 1 and 2 of each week under the supervision of licensed physical therapists. Participants will have the choice of using a treadmill or a recumbent stepper. The physical therapists will monitor blood glucose level, blood pressure, heart rate, and RPE during each exercise session. Participants will be asked to exercise at home on Day 3 of each week, and will not be supervised by the study team.

SUMMARY:
A pilot longitudinal study to examine hyaluronan (HA) accumulation in muscles of individuals with Type 2 diabetes mellitus (T2DM), and the effects of exercise on HA accumulation, muscle stiffness, strength, ankle joint mobility, and physical function. HA accumulation will be assessed non- invasively using magnetic resonance imaging.

DETAILED DESCRIPTION:
This single-center, longitudinal design study uses MRI to evaluate the mechanistic effects of exercise on skeletal muscle function. Twenty-five T2DM patients will be enrolled and be prescribed a 10-week exercise program. The exercise program will comprise aerobic and resistance components; a moderate level of intensity will be calculated based on results from a maximal graded exercise test (VO2R) conducted prior to the intervention. MRI data will be acquired at baseline and before and after the intervention that can provide mechanistic insight into the adaptations in lower leg muscle function.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 40 and 75
* Clinical diagnosis of Type 2 diabetes
* Have a BMI less than 40 kg/m2 (due to magnet bore restrictions)
* Able to walk unassisted

Exclusion Criteria:

* Serious cardiac pathology or musculoskeletal problems that would limit exercise ability
* Current open wound or history of plantar ulcer for the last 3 months
* Partial foot amputations
* Inability to ambulate without assistive device
* Stroke or other central nervous system pathology
* Stage 2 hypertension (resting blood pressure >160 systolic or >100 diastolic)
* Contraindications to 3T whole body MRI scanners (e.g., pacemaker, cerebral aneurysm clip, cochlear implant, presence of shrapnel in strategic locations, metal in the eye, claustrophobia, or other problems).
* Subjects with alcoholism, chronic drug use, chronic gastrointestinal disease, or renal or hepatic impairment
* Pregnant women and children

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the Level of Hyaluronan accumulation in calf muscle of participants | Week 1, Week 11
  Hyaluronan accumulation (HA) in calf muscle will be assessed using 3D T1ρ and T2-weighted MR scans on a 3T whole-body clinical MRI scanner (Prisma, Siemens Healthcare, Erlangen, Germany) with a 15-channel knee coil (QED, Cleveland OH). The total scan time is expected to be 29 min, 30 s. The sequence acquisition parameters will be as follows: TR/TE = 1500 ms/3.78 ms, flip angle = 8°, field of view (FOV) = 140 mm2, spin-lock lengths (TSLs)=0,10ms, 20ms, 30ms, 40ms and 60ms, spin-lock frequency=500Hz matrix size 256 × 128 × 64, slice thickness = 2 m.
Change in the Level of Calf muscle stiffness in participants | Week 1, Week 11
  Calf muscle stiffness will measured using a previously validated device (FDA product classification: non-powered goniometer, 510K exempt). Brieﬂy, subjects are positioned supine with the knee extended and their leg is secured by Velcro straps. Torques of 15, 20 and 25 Nm are applied using a hand-held force gauge (FDK 40, Wagner Instruments, Greenwich, CT) and resultant angular kinematics are measured using a digital inclinometer (Checkpoint Inc., Torrance, CA). Three cycles of testing are performed in ascending order of force application and resultant peak dorsiﬂexion range of motion is recorded at each force level. Calf muscle stiffness is calculated as the slope of the resultant curves over the 15 to 25 Nm intervals. This device has demonstrated high convergent validity compared to motion analysis (Intraclass correlation coefficient (ICC [2,k])> 0.95).
Change in the Degree of Passive ankle mobility in participants | Week 1, Week 11
  Passive ankle mobility will measured using a previously validated device (FDA product classification: non-powered goniometer, 510K exempt). Brieﬂy, subjects are positioned supine with the knee extended and their leg is secured by Velcro straps. The axis of rotation of the device is then adjusted in the anteroposterior and supero-inferior directions to approximate the ankle axis of rotation determined by palpation of the distal tips of the medial and lateral malleoli. Torques of 15, 20 and 25 Nm are applied using a hand-held force gauge (FDK 40, Wagner Instruments, Greenwich, CT) and resultant angular kinematics are measured using a digital inclinometer (Checkpoint Inc., Torrance, CA). Three cycles of testing are performed in ascending order of force application and resultant peak dorsiflexion range of motion is recorded at each force level.
Change in the Level of Calf muscle strength in participants | Week 1, Week 11
  Calf muscle strength, quantified as peak plantarflexion torque. An isokinetic dynamometer (Biodex, Shirley, NY) will be used to quantify peak isokinetic torque of the calf muscle at 60 degrees per second in participants' available range of motion (FDA product classification: AC powered dynamometer, 510K exempt). All participants will be tested in the seated position. Three practice trials will be given, after which peak plantarflexion torque will be recorded from the highest of three trials. With these procedures, coefficient of variation of <10% has been reported in individuals with T2DM, indicating good repeatability.
Change in the Change in Gait (Stride length) of participants after intervention | Week 1, Week 11
  The study will use a motion capture system to collect kinematic (marker) and kinetic (force plate and pressure plate) data as subjects walk barefoot at self-selected speed along a 10 m walkway. A minimum of five successful trials will be collected for each subject. A trial will be considered successful if the subject made clean force plate contact on the tested side without targeting. Stride length will be defined as the distance between consecutive initial contacts of the same limb and will be calculated using Visual3D software (C-motion Inc., USA).
Change in the Change in Gait (Walking Speed) of participants after intervention | Week 1, Week 11
  The study will use a motion capture system to collect kinematic (marker) and kinetic (force plate and pressure plate) data as subjects walk barefoot at self-selected speed along a 10 m walkway. A minimum of five successful trials will be collected for each subject. A trial will be considered successful if the subject made clean force plate contact on the tested side without targeting. Walking speed will be defined as distance travelled in unit time and will be calculated using Visual3D software (C-motion Inc., USA).
Change in Self-reported physical function of participants after intervention | Week 1, Week 11
  This will be evaluated using Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function and Pain Interference scales. PROMIS is a computer adaptive testing outcomes instrument, generated after exhaustive review, and the application of item response theory to calibrate the individual items. The higher the score indicate higher levels of physical functioning. All PROMIS measures are scored using the final re-centered item response theory (IRT) item parameters and transformed to the T-score metric (mean=50, SD=10).

SECONDARY OUTCOMES:
Change in the Glycemic Control | Week 2, Week 12
  Glycemic control will be assessed with Hemoglobin A1c test. Participants will be asked to give 1 mL of blood at baseline and after intervention.
Change in the Number of participants with increased physical activity | Week 1, Week 11
  Physical activity will be assessed using a wrist-worn triaxial accelerometer (Actigraph). Step counts, and percent of time in sedentary, light and moderate / vigorous physical activity will be quantified for each participant. The actigraph will be worn for two weeks on the wrist, participants may take it off when bathing and sleeping.
Number of Participants who adhere to the Exercise program | Week 12
  Number of sessions attended will be calculated and used to calculate adherence. A systematic review of exercise training indicates attrition rates of <20% and adherence rates of >75% in individuals with T2DM.
Number of participants with Neuropathy | Week 1
  The Michigan Neuropathy Screening Instrument will be used to screen for the presence of peripheral neuropathy. The Michigan Neuropathy Screening Instrument (MNSI) is used to assess distal symmetrical peripheral neuropathy in diabetes. It includes two separate assessments: a 15-item self-administered questionnaire and a lower extremity examination that includes inspection and assessment of vibratory sensation and ankle reflexes
Number of participants with Osteoarthritis | Week 1
  Presence of knee osteoarthritis may affect levels of serum HA. American College of Rheumatology (ACR) Clinical Classification Criteria will be used to screen for the presence of knee osteoarthritis. History and physical examination will be used to screen for knee osteoarthritis using the following criteria: Pain in the knee and three of the following: 1) >50 years of age, 2) Less than 30 minutes of morning stiffness, 3) Crepitus on active motion, 4) Bony tenderness, 5) Bony enlargement, 6) No palpable warmth of synovium.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Rao, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Available after accepted for publication in a peer-reviewed journal.
Access Criteria: Requests should be directed to smita.rao@nyu.edu. To gain access, data requestors will need to sign a data access agreement.